CLINICAL TRIAL: NCT04388007
Title: Predictors for Identifying Patients With Non-specific Back Pain Who Respond Favorably to Spinal Manipulation: a Prospective Cohort Study
Brief Title: Non-specific Back Pain and Spinal Manipulation
Status: Completed | Type: Observational
Sponsor: Université du Québec à Trois-Rivières (Other)
Responsible Party: Principal Investigator, Martin Descarreaux, Professor, Doctor of Chiropractic, Université du Québec à Trois-Rivières
Other Study IDs: UQTR-2020-SMTdose
Record Dates: First submitted 2020-05-07; First posted 2020-05-14 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Non-specific Back Pain
Keywords: Back pain; Spinal manipulation; Cohort study
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Thoracic spinal manipulation — High velocity, low amplitude force manipulation

SUMMARY:
The main purpose of this study is to identify short-term predictors of positive responses to a spinal manipulation treatment. To do this, positive responses to treatment, characterized by improvement in pain score, functional capacity, as well as the global perceived change will be evaluated using single and multiple logistic regressions in which biomechanical variables, comfort, expectation will used as potential predictors.

DETAILED DESCRIPTION:
The main purpose of this study is to identify short-term predictors of positive responses to a spinal manipulation treatment. To do this, positive responses to treatment, characterized by improvement in pain score, functional capacity, as well as the global perceived change will be evaluated at baseline and at 7 days. Pain score will be also assessed every day with text-tracking. Global perceived change will be evaluated using single and multiple logistic regressions in which biomechanical variables, comfort, expectation will used as potential predictors. 100 individuals with a history of non-specific back pain will be recruited in a chiropractic care center.

ELIGIBILITY:
Inclusion Criteria:

* Being aged over 18 years old
* Presenting non-specific back pain (chronic >=3 months or recurrent complaint)
* Speaking French or English

Exclusion Criteria:

* Symptomatic thoracic pain
* Non-musculoskeletal disorders pain
* Pregnancy
* Not eligible to spinal manipulation (if osteoporosis, vertebral fracture history, thoracic disk herniation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants are patient in the chiropractic care center
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Thoracic Back Pain (Numerical Analog Scale) | change from baseline to Day-7
  assessed by a 0-10 points scale, higher score means altered, lower score means improved
Functional Disability (Quebec Back Pain Disability Scale) | change from baseline to Day-7
  assessed by 0-100 points questionary. Higher scores correlate to greater disability
Global Perceived Change Scale | at day-7
  assessed by a 11-point score scale: higher score means improved, lower score means altered

SECONDARY OUTCOMES:
Dosage | during the intervention
  assessed by a force-sensing table recording data through a computer software
Expectation (for improvement of pain and disability) | at baseline (pre-intervention)
  assessed by a 11-point score scale : higher score means improved, lower score means altered
Socio-demographic factors | at baseline(pre-intervention)
  assessed with a patient history questionary
Tampa Scale of Kinesiophobia | at baseline(pre-intervention)
  Questionary, Total score range from 17 to 68, Higher score indicate a worst outcome
Level of anxiety | at baseline (pre-intervention)
  Assessed using the State-Trait Anxiety Inventory (STAI) (score range from 20 (minimum) to 80 (maximum) : higher score mean a worst outcome)
Level of Comfort | at baseline (post-intervention)
  Assessed with a 100mm scale : higher score means very comfortable

CONTACTS AND LOCATIONS:
Overall Officials: Martin Descarreaux, DC, PhD, Study Director — Université du Québec à Trois-Rivières
Locations (1):
- Université du Québec à Trois-Rivières, Trois-Rivières, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No